CLINICAL TRIAL: NCT00823979
Title: A Phase 2b Multicenter, Randomized, Comparative Trial Of Uk-453,061 Versus Etravirine In Combination With Darunavir/Ritonavir And A Nucleotide/Nucleoside Reverse Transcriptase Inhibitor For The Treatment Of Antiretroviral Experienced Hiv-1 Infected Subjects With Evidence Of Nnrti Resistant Hiv-1
Brief Title: A Phase 2B Multicenter, Randomized, Comparative Trial Of UK-453,061 Versus Etravirine In Combination With Darunavir/Ritonavir And A Nucleos(t)Ide Reverse Transcriptase Inhibitor For The Treatment Of Antiretroviral Experienced HIV-1 Infected Subjects With Evidence Of NNRTI Resistant HIV-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5271022; 2007-004392-19 (EudraCT Number)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: HIV-1
Keywords: HIV-1 NNRTI Treatment Experienced; may have Protease inhibitor experience
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UK- 453,061 Dose One (Experimental)
  Interventions: Drug: UK-453,061 Dose 1
- UK- 453,061 Dose Two (Experimental)
  Interventions: Drug: UK-453,061 Dose 2
- Comparator (Active Comparator)
  Interventions: Drug: Etravirine

INTERVENTIONS:
Drug: UK-453,061 Dose 1 — UK 453,061 750 mg QD + one optimized NRTI + darunavir/ritonavir.
  Arms: UK- 453,061 Dose One
Drug: UK-453,061 Dose 2 — UK 453,061 1000 mg QD + one optimized NRTI + darunavir/ritonavir.
  Arms: UK- 453,061 Dose Two
Drug: Etravirine — Etravirine 200 mg BID + one optimized NRTI + darunavir/ritonavir.
  Arms: Comparator

SUMMARY:
This is a 96 week study to determine if UK- 453,061 in combination with Darunavir /ritonavir and a Nucleos(t)ide Reverse Transcriptase inhibitor is as efficacious, safe and tolerable as etravirine in combination with Darunavir /ritonavir and a Nucleos(t)ide Reverse Transcriptase inhibitor in HIV-1 infected patients who have been previously treated with antiretroviral drugs and have NNRTI resistance mutations.

DETAILED DESCRIPTION:
The trial was terminated on 12 April, 2012 due to lack of efficacy at the Week 24 analysis. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age available for a follow-up period of at least 96 weeks.
* HIV 1 RNA viral load of greater then 500 copies/mL.
* Negative urine pregnancy test.

Exclusion Criteria:

* Suspected or documented active, untreated HIV-1 related opportunistic infection or other condition requiring acute therapy at the time of randomization.
* Subjects with acute Hepatitis B and/or C within 30 days of randomization.
* Previous use of Darunavir or etravirine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2012-10-18 (Actual); Study Completion 2012-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (21):
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Office of Anthony Mills, MD, Inc., Los Angeles, California
  - CARES, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - The Kinder Medical Group, Miami, Florida
  - Care Resource, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Diseases Associates of Northwest Florida, PA, Pensacola, Florida
  - Hillsborough County Health Department, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Nassau University Medical Center, East Meadow, New York
  - Greiger Clinic, Mount Vernon, New York
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Saint Hope Foundation - Bellaire Clinic, Bellaire, Texas
  - Saint Hope Foundation - Conroe Clinic, Conroe, Texas
  - Nicholaos C. Bellos, MD, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Saint Hope Foundation - Stafford Clinic, Stafford, Texas
- Brazil (6):
  - Instituto A.Z. de Pesquisa e Ensino, Curitiba, Paraná
  - Hospital Geral de Nova Iguacu, Nova Iguaçu, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto de Infectologia Campinas, Campinas, São Paulo
  - Centro de Referencia e Treinamento DST/AIDS, São Paulo, São Paulo
  - Hospital Heliopolis, São Paulo, São Paulo
- Klinikum der Universitaet zu Koeln, Klinik I fuer Innere Medizin, Cologne, Germany
- Italy (2):
  - Unita' Operativa Malattie Infettive, Bologna
  - U.O.S. Immunologia Clinica, Roma
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur
- Poland (2):
  - Oddzial do Leczenia HIV, Szczecin
  - SPZOZ Wojewodzki Szpital Zakazny, Warsaw
- Portugal (5):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa - Zona Central - Hospital Santo António Capuchos, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE., Lisbon
  - Hospital São João, Porto
  - Hospital de Joaquim Urbano, Porto
- Puerto Rico (5):
  - UPR-CTU Pharmacy, San Juan, PR
  - Innovative Care PSC, Bayamón
  - Ararat Research Center, Ponce
  - University of Puerto Rico - Medical Sciences Campus - Puerto Rico Medical Center, Rio Piedras
  - HOPE Clinical Research, San Juan
- South Africa (7):
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - University of Witwatersrand, Johannesburg, Gauteng
  - Chris Hani Baragwanath Hospital, Soweto, Johannesburg
  - Dr. J Fourie Medical Centre, Dundee, KwaZulu-Natal
  - 203 Maxwell Centre, Durban, KwaZulu-Natal
  - Willowmead Medical Center, Cape Town, Western Cape
  - Desmond Tutu HIV Foundation, Cape Town, Western Cape
- Spain (2):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitario La Paz, Madrid
- Taiwan (2):
  - Department of Infectious Disease, E-Da Hospital, Kaohsiung County
  - Veterans General Hospital - Taipei, Taipei
- Ukraine (3):
  - Vinnitsa Regional center for AIDS Prevention and Control, Berezyna, Vinnitsa District, Vinnitsa Region
  - Donetsk Regional Center of AIDSs prophylaxis and control, Donetsk
  - Lugansk Regional Center of AIDS prophylaxis and control, Luhansk
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, EAST Sussex
  - North Manchester General Hospital, Crumpsall, Greater Manchester
  - Royal Infirmary GUM Clinic, Edinburgh
  - Western General Hospital, Edinburgh
  - Royal Free Hospital, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Lersivirine 750 mg: Lersivirine (UK-453,061) 250 milligram (mg) 3 tablets equivalent to lersivirine 750 mg and 1 placebo tablet matched to lersivirine 250 mg tablet, orally once daily up to 96 weeks in combination with 1 optimized nucleoside reverse transcriptase inhibitors (NRTI) as per individual prescribing information, darunavir 600 mg tablet orally twice daily and ritonavir 100 mg tablet or capsule orally twice daily.
- Lersivirine 1000 mg: Lersivirine (UK-453,061) 250 mg 4 tablets equivalent to lersivirine 1000 mg, orally once daily up to 96 weeks in combination with 1 optimized NRTI as per individual prescribing information, darunavir 600 mg tablet orally twice daily and ritonavir 100 mg tablet or capsule orally twice daily.
- Etravirine 200 mg: Etravirine 100 mg 2 tablets equivalent to etravirine 200 mg, orally twice daily up to 96 weeks in combination with 1 optimized NRTI as per individual prescribing information, darunavir 600 mg tablet orally twice daily and ritonavir 100 mg tablet or capsule orally twice daily.
Period: Overall Study
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Started | 35 | 35 | 35
Treated | 31 | 32 | 34
Completed | 6 | 3 | 11
Not Completed | 29 | 32 | 24
Not completed — Lack of Efficacy | 13 | 16 | 9
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 4
Not completed — Other | 2 | 0 | 1
Not completed — Randomized but not Treated | 4 | 3 | 1
Not completed — Study Terminated by Sponsor | 5 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg | Total
Number analyzed (Participants) | 31 | 32 | 34 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (8.9) | 40.0 (8.7) | 41.9 (9.1) | 41.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 18 | 51
  Male | 16 | 14 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus Type 1 Ribonucleic Acid (HIV-1 RNA) Levels Less Than (<) 50 Copies/Milliliter (mL) at Week 24
Description: Plasma HIV-1 RNA level was determined by the Roche Amplicor HIV-1 Monitor standard assay (version 1.5).
Time Frame: Week 24
Population: ITT population. Participants who died, discontinued, lost to follow-up, switched/changed dose of anti-retro viral (ARV) drug not allowed by protocol, had missing plasma HIV-1 RNA data at 24 weeks were considered to have plasma HIV-1 RNA >=50 copies/mL and were referred to as failure.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
percentage of participants | 48.4 | 43.8 | 67.6

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels <50 Copies/mL at Week 48 and 96
Description: Plasma HIV-1 RNA level was determined by the Roche Amplicor HIV-1 Monitor standard assay (version 1.5).
Time Frame: Weeks 48, 96
Population: ITT population. Participants who died, discontinued,lost to follow-up,switched/changed dose of ARV drug not allowed by protocol,had missing plasma HIV-1 RNA data at 48, 96 weeks were considered to have plasma HIV-1 RNA >=50 copies/mL and were referred to as failure. n=participants evaluable at specified time point for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
percentage of participants
  Week 48 (n=31, 32, 34) | 41.9 | 31.3 | 61.8
  Week 96 (n=28, 28, 27) | 25.0 | 14.3 | 37.0

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels <400 Copies/mL at Week 24, 48 and 96
Description: Plasma HIV-1 RNA level was determined by the Roche Amplicor HIV-1 Monitor standard assay (version 1.5).
Time Frame: Week 24, 48, 96
Population: ITT population. Participants who died,discontinued,lost to follow-up,switched/changed dose of ARV drug not allowed by protocol,had missing plasma HIV-1 RNA data at 24, 48, 96 weeks were considered to have plasma HIV-1 RNA >=400 copies/mL and referred to as failure. n=participants evaluable at specified time point for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
percentage of participants
  Week 24 (n=31, 32, 34) | 54.8 | 50.0 | 79.4
  Week 48 (n=31, 32, 34) | 41.9 | 34.4 | 70.6
  Week 96 (n=28, 28, 27) | 25.0 | 14.3 | 37.0

4. Secondary Outcome: Change From Baseline in log10 Transformed HIV-1 RNA Levels at Week 24, 48 and 96
Description: Plasma HIV-1 RNA level was determined by the Roche Amplicor HIV-1 Monitor standard assay (version 1.5). For the log10 scale, all the HIV-1 RNA levels were log10 transformed prior to the average calculations. Baseline value calculated as average of measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline, Week 24, 48, 96
Population: ITT population. Participant discontinued before a visit of interest: value imputed as zero; not discontinued but observation is missing: last observation carried forward (LOCF) imputation used; missing baseline or no HIV-1 RNA level assessment: value imputed as zero.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
log10 copies/mL
  Baseline | 4.28 (0.99) | 4.76 (0.82) | 4.59 (0.79)
  Change at Week 24 | -1.53 (1.58) | -1.89 (1.46) | -2.32 (1.21)
  Change at Week 48 | -1.30 (1.64) | -1.08 (1.48) | -2.06 (1.42)
  Change at Week 96 | -0.69 (1.39) | -0.36 (1.00) | -0.96 (1.49)

5. Secondary Outcome: Time-Averaged Difference (TAD) in log10 Transformed HIV-1 RNA Levels at Week 24, 48 and 96
Description: TAD was calculated as (area under the curve of HIV-1 RNA levels [log10 copies/mL] from baseline to the time point of interest divided by time period in weeks) minus baseline HIV-1 RNA level (log10 copies/mL). Baseline value calculated as average of measurements collected at prior to and including Day 1 pre-dose. Due to early termination of the study decision was made not to derive TAD results for Week 96.
Time Frame: Week 24, 48, 96
Population: ITT population. Participant discontinued before a visit of interest: TAD imputed as zero; not discontinued but observation was missing at visit: TAD to the last non-missing timepoint; not discontinued and missing values between baseline and visit: ignore missing values; missing baseline or no HIV-1 RNA level assessment: TAD imputed as zero.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
log10 copies/mL
  Week 24 | -1.46 (1.12) | -1.72 (1.11) | -2.10 (0.92)
  Week 48 | -1.28 (1.39) | -1.19 (1.35) | -1.89 (1.27)

6. Secondary Outcome: Percentage of Participants With Response as Determined by the Time to Loss of Virologic Response (TLOVR50) Algorithm at Week 24, 48 and 96
Description: TLOVR50 response (50 denotes lower limit of quantification [LLOQ] of assay=50 copies/mL): compliment to TLOVR50 failure. TLOVR50 failure based on observed HIV-1 RNA levels and failure events (death; permanent discontinuation of drug; lost to follow-up; new ARV drug; met treatment failure [TF] criteria). TF: an increase of at least (>=)3 times the baseline plasma HIV-1 RNA level at Week 2 or thereafter; failure to achieve HIV-1 RNA level <50 copies/mL at Week 24; starting at Week 2, an increase in HIV-1 RNA level to detectable levels (>50 copies/mL); HIV-1 RNA <1 log10 decrease from baseline at Week 4 or thereafter. TF were confirmed by second measurement >=14 days after first. Baseline value was calculated as the average of the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Week 24, 48, 96
Population: ITT.Participants who died,discontinued,lost to follow-up,switched/changed dose of ARV drug not allowed by protocol,had missing plasma HIV-1 RNA data at 24,48 weeks were considered to have plasma HIV-1 RNA>=50 copies/mL;were referred as failure. Due to early termination of study,decision was made not to derive TLOVR50 responder analysis for Week 96.
Measure: Number; unit: percentage of participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
percentage of participants
  Week 24 | 48.4 | 43.8 | 67.6
  Week 48 | 41.9 | 28.1 | 55.9

7. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Absolute Lymphocyte Counts at Week 24, 48 and 96
Description: Blood samples for immunological status assessed by CD4+ lymphocyte count. Baseline value was calculated as the average of the measurements collected prior to and including Day 1 pre-dose.
Time Frame: Baseline, Week 24, 48, 96
Population: ITT population included all randomized participants who received at least 1 dose of study drug. Missing values were imputed using LOCF. Participants with missing baseline or no CD4+ count available on treatment imputed as no or zero change from baseline.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/mcL)
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
cells per microliter (cells/mcL)
  Baseline | 247 (143) | 259 (187) | 227 (146)
  Change at Week 24 | 98 (140) | 66 (111) | 110 (108)
  Change at Week 48 | 122 (148) | 74 (128) | 128 (127)
  Change at Week 96 | 148 (177) | 89 (152) | 184 (197)

8. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Percentage Lymphocyte Counts at Week 24, 48, 96
Description: as for outcome 7
Time Frame: Baseline, Week 24, 48, 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of total lymphocytes
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 31 | 32 | 34
percentage of total lymphocytes
  Baseline | 16.1 (8.7) | 15.0 (8.8) | 14.6 (8.3)
  Change at Week 24 | 3.0 (4.0) | 3.7 (3.6) | 3.7 (3.2)
  Change at Week 48 | 4.6 (5.3) | 4.0 (4.1) | 4.4 (3.8)
  Change at Week 96 | 5.4 (6.1) | 4.2 (4.9) | 6.2 (6.2)

9. Secondary Outcome: Number of Participants With Non-nucleoside Reverse Transcriptase Inhibitors (NNRTI) Resistance-Associated Mutations (RAMs) and/or Phenotypic Susceptibility at Time of Treatment Failure Through Week 48
Description: Genotypic and phenotypic resistance to NNRTIs based on International Acquired Immunodeficiency Syndrome (AIDS) Society, United States of America (IAS-USA) RAM guidelines were evaluated using Monogram Biosciences PhenoSenseGT Assay at Baseline. This was then repeated for all participants with HIV-1 viral load >500 copies/mL at treatment failure, up to Week 48.
Time Frame: Baseline through Week 48
Population: Virology analysis set included a subset of participants from TLOVR50 failures who had valid genotypic or phenotypic susceptibility testing result and with plasma HIV-1 RNA >500 copies/mL at baseline and treatment failure.
Measure: Number; unit: participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 12 | 16 | 4
participants | 5 | 3 | 1

10. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory analysis included blood chemistry, hematology and urinalysis.
Time Frame: Baseline up to Week 48 or early termination
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 29 | 31 | 34
participants | 27 | 30 | 33

11. Secondary Outcome: Population Pharmacokinetics (PK) of Lersivirine
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48
Reporting Status: Not Posted

12. Secondary Outcome: Lersivirine Success Percentage With Reference to Median Minimum Observed Plasma Concentration (Cmin)
Description: Simple quartile exposure analysis of success rate (viral load <50 copies/mL) versus median Cmin assesses the exposure response relationship. Percentage of participants with HIV-1 RNA level <50 copies/mL at median Cmin quartile were planned to be reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48
Population: Due to the sparsity of the data, the ability to interpret the pharmacokinetic/pharmacodynamic (PK/PD) results was limited, thus the data was not reported.
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Lersivirine 750 mg | Lersivirine 1000 mg | Etravirine 200 mg
Serious Adverse Events (participants affected / at risk) | 1/31 | 4/32 | 1/34
Other Adverse Events (participants affected / at risk) | 27/31 | 25/32 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine 750 mg (N=31) | Lersivirine 1000 mg (N=32) | Etravirine 200 mg (N=34)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine 750 mg (N=31) | Lersivirine 1000 mg (N=32) | Etravirine 200 mg (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 7 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 14 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 3
Asthenia (General disorders) | 0 | 1 | 0
Fat tissue increased (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 0
Body tinea (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2
Dermatophytosis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 5
Hordeolum (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 4 | 0 | 4
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Myringitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral hairy leukoplakia (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Papilloma viral infection (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 2 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Trichomoniasis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radiation associated pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Tetrahydrocortisol urine increased (Investigations) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1
Headache (Nervous system disorders) | 2 | 2 | 4
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypogeusia (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Arterial spasm (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated on 12 April, 2012 due to lack of efficacy at the Week 24 analysis. The decision to terminate the trial was not based on any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.